CLINICAL TRIAL: NCT01119560
Title: Genetic Susceptibility Factors in the Etiology of Neuroblastoma Also Known as Neuroblastoma Epidemiology in North America (NENA)
Brief Title: Genetic Susceptibility Biomarkers in Children With Neuroblastoma (Also Known as Neuroblastoma Epidemiology in North America [NENA])
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AEPI07N1; NCI-2011-02257 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-AEPI07N1; CDR0000594334; AEPI07N1 (Other: Childrens Oncology Group); AEPI07N1 (Other: CTEP); U10CA180886 (NIH); U10CA098543 (NIH)
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

GROUPS / COHORTS (1):
- Ancillary-Correlative (Questionnaire, saliva & tissue sample): The biologic mother of the patient is asked to complete a Diet History Questionnaire about diet during pregnancy, and information on demographics, lifestyle factors, medication used during pregnancy, history of breast feeding, and family history of cancer or birth defects. Parents are given ORAgene saliva collection kits for self-collection. Saliva bio-specimen samples are collected from both biologic parents and the patient. Tissue samples previously stored in a tissue bank are obtained for deceased patients, if available. DNA is extracted from samples, amplified and analyzed using real-time PCR quantitation assay, and genotyped using single nucleotide polymorphisms.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Correlative studies
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This research trial studies the genes biomarkers in children with neuroblastoma. Studying the genes in a child's cancer cells may help doctors improve ways to diagnose and treat children with neuroblastoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the independent association of common genetic polymorphisms involved in folate, vitamin A, and related metabolic and transport pathways and the risk of neuroblastoma (NB).

II. Evaluate the joint effects of multiple genes on the risk of NB. III. Evaluate the effects of gene-exposure interactions on the risk of NB. IV. Evaluate genetic effects within NB subgroups defined by age at diagnosis and a Children?s Oncology group classification schema based on age, v-myc avian myelocytomatosis viral oncogene neuroblastoma derived homolog (MYCN) oncogene status, histology, and deoxyribonucleic acid (DNA) ploidy.

V. Recontact mothers of participating NENA case children, conduct brief web-based screen to ascertain whether the pregnancy including the index NENA child was a multiple (twin, triplet, etc), whether the mother knew if the children were monozygotic (MZ) or dizygotic (DZ), and obtain a complete pregnancy history.

VI. Request a saliva sample from the other twin/multiple sibling of the NENA child.

VII. Extract DNA from saliva samples and securely store. VIII. Clean new survey data and merge with main NENA study database.

OUTLINE:

The biologic mother of the patient is asked to complete a Diet History Questionnaire about diet during pregnancy, and information on demographics, lifestyle factors, medication used during pregnancy, history of breast feeding, and family history of cancer or birth defects. Parents are given ORAgene saliva collection kits for self-collection. Saliva bio-specimen samples are collected from both biologic parents and the patient. Tissue samples previously stored in a tissue bank are obtained for deceased patients, if available. DNA is extracted from samples, amplified and analyzed using real-time polymerase chain reaction (PCR) quantitation assay, and genotyped using single nucleotide polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of neuroblastoma made at a North American COG institution
* Diagnosed between 12/24/2007- 7/31/2013
* Diagnosed at < 6 years of age
* Biological mother is alive and willing to participate
* Questionnaire respondents must understand English or Spanish
* Are only those participating in CCRN who have agreed to be contacted for future studies

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Sampling Method: Probability Sample
Enrollment: 576 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Genetic polymorphisms involved in folate, vitamin A, and related metabolic and transport pathways with the risk of neuroblastoma (NB) | Up to 4 years
  The distributions of the estimated dietary and vitamin intake will be assessed and categories defined using quantiles and confirmation by nonparametric splines. Evaluated under a recessive or log-additive transmission model.
Gene-exposure interactions, with primary interest on folate, vitamin A, and choline intake, on the risk of NB | Up to 4 years
  Stratified on the exposure variable and the strength of associations between strata by using a chi-square based test of heterogeneity.
Gene-environment interactions | Up to 4 years
  Stratified on the exposure variable and comparing the strength of associations between strata by using a chi-square-based test of heterogeneity.
Genetic effects within NB subgroups defined by age at diagnosis and a Children?s Oncology group classification schema based on age, MYCN oncogene status, histology, and deoxyribonucleic acid (DNA) ploidy | Up to 4 years
  Because the log-linear models involve calculating a likelihood, the Bayesian information criterion, a likelihood-based model selection criterion will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Olshan, Principal Investigator — Children's Oncology Group
Locations (153):
- United States (141):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - USA Health Strada Patient Care Center, Mobile, Alabama
  - Phoenix Childrens Hospital, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital Stanford University, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Rady Children's Hospital - San Diego, San Diego, California
  - UCSF Medical Center-Parnassus, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - University of Florida Health Science Center - Gainesville, Gainesville, Florida
  - Memorial Regional Hospital/Joe DiMaggio Children's Hospital, Hollywood, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - Miami Cancer Institute, Miami, Florida
  - Florida Hospital Orlando, Orlando, Florida
  - UF Cancer Center at Orlando Health, Orlando, Florida
  - Nemours Children's Clinic - Pensacola, Pensacola, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Hospital, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Egleston, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Lurie Children's Hospital-Chicago, Chicago, Illinois
  - University of Illinois, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital-Oak Lawn, Oak Lawn, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Ascension Saint John Hospital, Detroit, Michigan
  - Michigan State University Clinical Center, East Lansing, Michigan
  - Helen DeVos Children's Hospital at Spectrum Health, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital and Medical Center of Omaha, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Albany Medical Center, Albany, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - NYU Winthrop Hospital, Mineola, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University/Herbert Irving Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Mission Hospital Inc-Memorial Campus, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - East Carolina University, Greenville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Mercy Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Saint Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - BI-LO Charities Children's Cancer Center, Greenville, South Carolina
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center-Amarillo, Amarillo, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Vermont College of Medicine, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - British Columbia Children's Hospital, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Child Health Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Children's Hospital, London, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan